CLINICAL TRIAL: NCT00809705
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Investigate the Effect of Taspoglutide on Gastric Emptying Measured by a Paracetamol Test After Single Dose and After Multiple Doses in Patients With Type 2 Diabetes
Brief Title: A Study of the Effect of Taspoglutide on Gastric Emptying in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP21572; 2008-003575-47
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: taspoglutide
- 2 (Experimental)
  Interventions: Drug: taspoglutide
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — sc once weekly for 12 weeks
  Arms: 3
Drug: taspoglutide — 10mg sc once weekly for 4 weeks, followed by 20mg sc once weekly for 8 weeks
  Arms: 2
Drug: taspoglutide — 10mg sc once weekly for 12 weeks
  Arms: 1

SUMMARY:
This 3 arm, placebo-controlled study will investigate the effect of Taspoglutide on gastric emptying in patients with type 2 diabetes. Patients will be randomized into one of 3 groups to receive a)10mg Taspoglutide sc weekly for 12 weeks b)10mg Taspoglutide sc weekly for 4 weeks followed by 20mg Taspoglutide sc weekly for 8 weeks or c) placebo sc weekly for 12 weeks, with all injections administered in the abdomen.Gastric emptying will be assessed by a paracetamol test at intervals during the study. The anticipated time on study treatment is 3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes mellitus, treated with stable oral antidiabetic drug therapy for >=3 months prior to screening;
* stable weight +/-10% for >=3 months before screening.

Exclusion Criteria:

* type 1 diabetes mellitus;
* acute gastrointestinal symptoms at screening and/or day -1;
* clinically relevant cardiovascular, bronchopulmonary, gastrointestinal or neurological disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Tmax, log (AUC), log(Cmax)of paracetamol | Days -1, 1, 5, 29, 33, 78 and 82

SECONDARY OUTCOMES:
Adverse events, laboratory parameters, vital signs | Throughout study
renal function (creatinine clearance, urine volume and electrolytes) | Throughout study
Multiple dose pharmacokinetics of Taspoglutide | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Germany (2):
  - Berlin
  - Neuss
- London, United Kingdom